CLINICAL TRIAL: NCT06658353
Title: Single-arm, Open, Multi-center Phase III Clinical Study to Assess the Safety and Effectiveness of VC004 in Patients With Localized Advanced/ Metastatic Solid Tumors
Brief Title: Phase III Clinical Study of VC004 in Patients With Localized Advanced/ Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu vcare pharmaceutical technology co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VC004-301
Record Dates: First submitted 2024-10-24; First posted 2024-10-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VC004 Capsules (Experimental)
  Interventions: Drug: VC004 Capsules

INTERVENTIONS:
Drug: VC004 Capsules — VC004 Capsules BID

SUMMARY:
This Study is a single arm, open label, multicenter phase III clinical trial to evaluate the safety and efficacy of VC004 in patients with locally advanced/metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or legal representatives are willing and able to sign ICF approved by the ethics committee before starting any screening procedures；
* Male or female, age ≥12 years old;

Exclusion Criteria:

* Patients have undergone major surgery within 4 weeks prior to the first dose or are expected to undergo major surgery during the trial (excluding vascular access establishment procedures, biopsy procedures);
* Adverse reactions caused by previous treatment have not recovered to ≤1 grade (evaluated by the investigator);
* Patients had been treated with a strong CYP3A inhibitor or inducer within 7 days prior to the first administration of the study drug.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: yuankai Shi, Principal Investigator — Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Hospital,Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China